CLINICAL TRIAL: NCT07291362
Title: Artificial Intelligence Model-Assisted Improvement of Pathologists' Performance in Clinical Diagnostic Tasks: A Multicenter, Prospective, Randomized Controlled Trial
Brief Title: AI-Assisted Pathologist Performance Improvement: A Multicenter, Prospective, Randomized Controlled Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NFEC-2025-653
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pathology Foundation Model
Keywords: Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assisted group (Experimental): Doctors in this group are required to use the AI pathology diagnostic model to assist their diagnoses. The AI pathology model will provide a predicted result for each case.
  Interventions: Other: AI pathology model
- Independent Diagnosis Group (Control Group) (Placebo Comparator): In this group, pathologists will independently diagnose each case based on their own clinical experience, and will record both their time to diagnosis and their diagnostic confidence.
  Interventions: Other: Control

INTERVENTIONS:
Other: AI pathology model — Doctors in this group are required to use the AI pathology model to assist their diagnoses. The AI pathology model will provide a predicted result for each case.
  Arms: AI-assisted group
Other: Control — Pathologists will independently diagnose each case based on their own clinical experience, and will record both their time to diagnosis and their diagnostic confidence.
  Arms: Independent Diagnosis Group (Control Group)

SUMMARY:
The investigators plan to conduct a multicenter, prospective, randomized controlled trial to systematically evaluate the added value of pathology-based AI models in the gastric cancer diagnostic workflow. The study will focus on comparing AI-assisted platform interpretation with conventional independent slide reading in terms of diagnostic accuracy (e.g., AUC), reading efficiency (e.g., comparison of time to diagnosis), quality of diagnostic reports, diagnostic confidence (Likert scale), and pathologists' satisfaction with the AI models. The investigators will also assess superiority for less-experienced (junior) pathologists and noninferiority for more-experienced (senior) pathologists. Successful completion of this project will provide high-level prospective evidence to support the standardized deployment, quality control, and broader application of pathology AI in the gastric cancer care pathway.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: ≥ 18 years of age;
2. Patients undergoing gastric mucosal biopsy or gastric cancer surgical resection, with available digital pathology images and clinical information.

Exclusion Criteria:

1.Missing data or data of insufficient quality for analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Area under ROC curve (AUC) | Assessments will be conducted within one week after the physicians' diagnoses.
  Area under the curve

SECONDARY OUTCOMES:
Diagnostic time per case | Measured immediately after the physician's diagnosis.
  Time required for the pathologist to complete the diagnosis of each case in the AI-assisted diagnosis group compared with the independent diagnosis group. Diagnostic time is defined as the duration (in minutes/seconds) from initiating case review to finalizing and submitting the diagnostic report in the study system
Diagnostic report quality score | Within 1 week after the initial diagnosis for each case.
  Quality score of pathology diagnostic reports in the AI-assisted diagnosis group compared with the independent diagnosis group. Report quality will be evaluated by an independent panel of expert pathologists using a predefined scoring rubric (e.g., 0-100 scale), considering diagnostic accuracy, completeness, clarity, and structure of the report. Higher scores indicate better report quality.
Pathologists' diagnostic confidence | At the time of diagnosis for each case.
  Self-reported diagnostic confidence of pathologists for each case in the AI-assisted diagnosis group compared with the independent diagnosis group. Diagnostic confidence will be rated by the reporting pathologist on a [5]-point Likert scale (e.g., 1 = very uncertain to 5 = very confident) immediately after completing the diagnosis. Higher scores indicate greater diagnostic confidence.
Pathologists' satisfaction with the AI pathology model | Assessed once at the end of the AI-assisted reading period for each pathologist.
  Overall satisfaction of pathologists with the AI pathology diagnostic model in terms of usability and perceived effectiveness. Satisfaction will be assessed using a structured questionnaire comprising Likert-scale items that evaluate ease of use, integration into workflow, clarity of AI outputs, perceived impact on diagnostic efficiency, and perceived impact on diagnostic accuracy and confidence. Higher scores indicate higher satisfaction, better usability, and greater perceived effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Li Liang, Study Director — Nanfang Hospital, Southern Medical University
Locations (2):
- China (2):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No